CLINICAL TRIAL: NCT03720483
Title: Pilot Study to Evaluate Inhaled N-Acetylcysteine in Pulmonary Fibrosis
Brief Title: Inhaled NAC in Treatment of IPF
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study encountered challenges during startup due to the COVID-19 epidemic and was withdrawn.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-1477
Record Dates: First submitted 2018-07-18; First posted 2018-10-25 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetyl cysteine then placebo (Experimental): This arm will receive NAC followed by placebo
  Interventions: Drug: N-acetyl cysteine then Placebo
- Placebo then N-acetyl cysteine (Experimental): This arm will receive placebo followed by NAC
  Interventions: Drug: Placebo then N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine then Placebo — Subject will receive N-acetyl cysteine first followed by Placebo
  Arms: N-acetyl cysteine then placebo
Drug: Placebo then N-acetyl cysteine — Subject will receive Placebo first followed by N-acetyl cysteine
  Arms: Placebo then N-acetyl cysteine

SUMMARY:
This study plans to learn more about the safety and tolerability of inhaled N-Acetylcysteine (NAC) in patients with pulmonary fibrosis. The study will also create a bank of data, blood, and sputum from IPF patients for future research.

DETAILED DESCRIPTION:
This study plans to learn more about the safety and tolerability of inhaled N-Acetylcysteine (NAC) in patients with pulmonary fibrosis. The study will also create a bank of data, blood, and sputum from IPF patients for future research.

NAC is a medication used to loosen thick mucus. NAC was initially licensed for use in 1968. It is on the World Health Organization's List of Essential Medicines, the most effective and safe medicines needed in a health system, and it is available as a generic medication and is not very expensive. Inhaled NAC has been used as a mucus-dissolving therapy in respiratory conditions with excessive and/or thick mucus production.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by study team with expertise in IPF utilizing standard ATS/ERS definition of "probable" or "definite" IPF
* DLCO >50% predicted
* FVC >60% predicted
* FEV1/FVC > 0.7

Exclusion Criteria:

* History of bronchospasm (requiring treatment)
* Current acute exacerbation of their IPF disease
* Current smoker
* Supplemental O2 requirement > 4 liters/min via nasal cannula
* History of asthma, COPD, coronary artery disease, or cancer
* Currently using NAC, hypertonic saline, or DNase (dornase alfa) inhalation therapy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Pulmonary function - FVC | Baseline, week 10, and week 18
  Measure changes in percent predicted FVC
Changes in Pulmonary function - DLCO | Baseline, week 10, and week 18
  Measure changes in percent predicted DLCO

CONTACTS AND LOCATIONS:
Overall Officials: Mark Steele, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No